CLINICAL TRIAL: NCT04128410
Title: A Study on Central Transport Characteristics of Flurbiprofen Axetil in Elderly Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Yi Feng, MD (Other)
Responsible Party: Sponsor-Investigator, Yi Feng, MD, Director of department of anesthesiology and painmanagement, Peking University People's Hospital
Organization: Peking University People's Hospital (Other)
Other Study IDs: 2019PHB169-01
Record Dates: First submitted 2019-10-14; First posted 2019-10-16 (Actual); Last update posted 2019-10-16 (Actual); Status verified 2019-10

CONDITIONS: Flurbiprofen Axetil; Cerebrospinal Fluid; Anesthesia, Spinal; Aged
Keywords: S-flurbiprofen, R-flurbiprofen; cerebrospinal fluid; aged

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (10):
- T1: At 5 minutes after flurbiprofen axetil injected intravenously, 7 aged patients' samples were required to be collected
- T2: At 10 minutes after flurbiprofen axetil injected intravenously, 7 aged patients' samples were required to be collected
- T3: At 15 minutes after flurbiprofen axetil injected intravenously, 7 aged patients' samples were required to be collected
- T4: At 20 minutes after flurbiprofen axetil injected intravenously, 7 aged patients' samples were required to be collected
- T5: At 25 minutes after flurbiprofen axetil injected intravenously, 7 aged patients' samples were required to be collected
- T6: At 30 minutes after flurbiprofen axetil injected intravenously, 14 patients' samples were required to be collected,including 7 younger patients
- T7: At 35 minutes after flurbiprofen axetil injected intravenously, 7 aged patients' samples were required to be collected
- T8: At 40 minutes after flurbiprofen axetil injected intravenously, 7 aged patients' samples were required to be collected
- T9: At 45 minutes after flurbiprofen axetil injected intravenously, 7 aged patients' samples were required to be collected
- T10: At 50 minutes after flurbiprofen axetil injected intravenously, 7 aged patients' samples were required to be collected

SUMMARY:
The project will apply the methods of clinical observation experiment to study the central transport characteristics of flurbiprofen axetil by detecting S-flurbiprofen and R-flurbiprofen concentrations in cerebral-spinal fluid(CSF) after intravenous injection of flurbiprofen axetil in elderly patients.

DETAILED DESCRIPTION:
The patients undergoing spinal anesthesia for lower extremity surgery will be studied. Flurbiprofen axetil 100mg will be injected intravenously. CSF 1ml and blood 2ml will be obtained simultaneously every 5 minutes after intravenous injection in 50 min( T1~T10).CSF and blood samples will be used to detected S-flurbiprofen and R-flurbiprofen concentrations by using Liquid Chromatography-Mass Spectrometry. And the CSF/blood S-flurbiprofen and R-flurbiprofen concentrations ratio were calculated.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing lower extremity surgery under spinal or combined spinal-epidural anesthesia will be selected.

Exclusion Criteria:

* asthma, liver insufficiency, renal insufficiency, peptic ulcer, allergy to NSAIDs, and a history use of NSAIDs within two weeks before operation.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: ASA I or lII, both sexes, aged 18-85 yr
Sampling Method: Non-Probability Sample
Enrollment: 77 (Estimated)
Dates: Start 2019-10 (Estimated); Primary Completion 2019-10 (Estimated); Study Completion 2019-10 (Estimated)

PRIMARY OUTCOMES:
The concentrations of S-flurbiprofen and R-flurbiprofen in plasma and CSF of all patients. | perioperation
  The samples will be used to be determined plasma and CSF drug concentrations.

CONTACTS AND LOCATIONS:
Overall Officials: Yi Feng, MD, Study Chair — Peking University People's Hospital
Locations (1):
- Peking University People's Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No